CLINICAL TRIAL: NCT04158050
Title: Comparison of Biologicals in Treatment of Severe Asthma - Real Life Experiences
Brief Title: Comparison of Biologicals in Treatment of Severe Asthma
Acronym: BiSA
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Ida Montini Foundation (Other)
Responsible Party: Principal Investigator, Paula Kauppi, MD, PhD, Chief Specialist of Allergy Department, Principal Investigator, Adj Prof., Helsinki University Central Hospital
Other Study IDs: HUS/25/2019
Record Dates: First submitted 2019-11-03; First posted 2019-11-08 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- anti-IL5/IL5R-therapy group: Asthma patients, asthma and rhinitis, asthma and nasal polyps and anti-IL5/IL5R
  Interventions: Drug: IL5 Antagonist or anti-IL5R-antibody or Omalizumab
- anti-IgE-therapy group: Asthma patients, asthma and rhinitis, asthma and nasal polyps and anti-IgE-therapy
  Interventions: Drug: IL5 Antagonist or anti-IL5R-antibody or Omalizumab

INTERVENTIONS:
Drug: IL5 Antagonist or anti-IL5R-antibody or Omalizumab — mepolizumab, reslizumab, benralizumab and omalizumab in severe asthma

SUMMARY:
This is a retrospective clinical study on adult patients (18 years or more) with biological therapy for severe asthma at the Helsinki University Central Hospital (HUCH). This is a real-life study with a broader patient population than in a randomized controlled trial. Omalizumab has been used for treatment of asthma in HUCH since January 2009, anti-IL5 therapies starting with mepolizumab since April 2016.

DETAILED DESCRIPTION:
The investigators collect and analyse results of anti-IL5/IL5R and anti-IgE therapies in asthma until October 2019.The investigators compare number of exacerbations, number of glucocorticoid courses, dose of per oral glucocorticoid, number of antibiotic courses, need of emergency care and hospitalizations because of asthma before use of biologicals and at the latest visits of the participants when using biologicals.

ELIGIBILITY:
Inclusion Criteria:

* asthma that remains uncontrolled despite moderate to high dose inhaled corticosteroid and additional therapy with at least one other controller medication and need for continuous per oral corticosteroids (OCS) or contraindications (or clinically significant side effects of OCS) against OCS and/or frequent courses (two or more per year) of OCS

Exclusion Criteria:

* patients without asthma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asthma patients that have received biologicals (anti-IL5/IL5R or anti-IgE) for asthma with or without chronic rhinitis and nasal polyps.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Kauppi, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kotisalmi E, Hakulinen A, Makela M, Toppila-Salmi S, Kauppi P. A comparison of biologicals in the treatment of adults with severe asthma - real-life experiences. Asthma Res Pract. 2020 May 13;6:2. doi: 10.1186/s40733-020-00055-9. eCollection 2020. PMID 32467765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
Started | 42 | 22 (This is a retrospective evaluation of clinical data)
Completed | 33 | 17
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group | Total
Number analyzed (Participants) | 42 | 22 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 21 | 55
  >=65 years | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9.75) | 48 (10.67) | 52 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 19 | 7 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 22 | 64
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 42 | 22 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Exacerbations of the Participants
Description: Change from the baseline in the number of courses of oral corticosteroids. Exacerbations of asthma estimated as number of courses of oral corticosteroids.
Time Frame: baseline (12 months before biologicals) and the latest (12 months after initiation of biologicals)
Measure: Mean (Standard Deviation); unit: Change in number of courses of oral c
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
Number analyzed (Participants) | 42 | 22
Change in number of courses of oral c | 2.77 (7.91) | 1.32 (2.01)

2. Secondary Outcome: Change in Oral Corticosteroid Dose in Milligrams
Description: Change in oral corticosteroid dose in milligrams
Time Frame: The baseline (at the time of the last outpatient before starting biologicals) and up to approximately 12 months for Anti-IL5/IL5R Therapy and approximately 44 months for the Anti-IgE Therapy"
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
Number analyzed (Participants) | 42 | 22
Milligrams | 3.0 (7.91) | 2.29 (5.80)

3. Secondary Outcome: Change in the Number of Courses of Antimicrobics
Description: Change in the number of courses of antimicrobics
Time Frame: The baseline (at 12 months before biologicals) and the latest 12 months after initiation of biologicals
Measure: Mean (Standard Deviation); unit: Change in antimicrobial courses/year
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
Number analyzed (Participants) | 42 | 22
Change in antimicrobial courses/year | 0.69 (2.08) | 0.23 (1.47)

4. Secondary Outcome: Change in the Number of Emergency Room Visits of the Participants
Description: Change in the number of emergency room visits of the participants
Time Frame: The baseline (at 12 months before biologicals) and the latest 12 months after initiation of biologicals
Measure: Mean (Standard Deviation); unit: Change in number of emergency visits
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
Number analyzed (Participants) | 42 | 22
Change in number of emergency visits | 0.29 (1.30) | 0.18 (1.19)

5. Other Pre Specified Outcome: Change in Number of Polypectomy, FESS and Ethmoidectomy
Description: Change in number of Polypectomy, FESS and ethmoidectomy
Time Frame: The baseline (before biologicals) and the latest 12 months after initiation of biologicals
Measure: Mean (Standard Deviation); unit: Procedures
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
Number analyzed (Participants) | 42 | 22
Procedures
  Polypectomy | 1.24 (3.03) | 1.41 (4.69)
  FESS | 0.95 (0.89) | 0.82 (1.25)
  Ethmoidectomy | 0.71 (0.94) | 0.12 (0.68)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the total time period in both treatment arms. The total treatment period for the anti-IL5/IL5R-therapy was a mean of 12.8 months (SD 8.5) and for the anti-IgE therapy a mean of 49.1 months (SD 35.3).
Description: Adverse events information was collected in the medical records.
Arm/Group | Anti-IL5/IL5R-therapy Group | Anti-IgE-therapy Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/22
Other Adverse Events (participants affected / at risk) | 7/42 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-IL5/IL5R-therapy Group (N=42) | Anti-IgE-therapy Group (N=22)
Pneumopleuritis and pericarditis (Cardiac disorders) | 1 (1) | 0 (0) — Pneumopleuritis and pericarditis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-IL5/IL5R-therapy Group (N=42) | Anti-IgE-therapy Group (N=22)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Fatique (Nervous system disorders) | 1 (1) | 1 (1)
Fever (Immune system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rise in transaminases (Gastrointestinal disorders) | 1 (1) | 0 (0)
Limb or joint pain or oedema (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Lip swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT04158050/Prot_SAP_000.pdf